CLINICAL TRIAL: NCT00134706
Title: A Phase II Study of Docetaxel Plus Carboplatin in Hormone Refractory Prostate Cancer Patients Refractory to Prior Docetaxel-based Chemotherapy
Brief Title: A Study of Docetaxel Plus Carboplatin in Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Beth Israel Deaconess Medical Center (Other); Lowell General Hospital (Other); Massachusetts General Hospital (Other); Oregon Health and Science University (Other); Wentworth-Douglass Hospital (Other)
Responsible Party: Mary-Ellen Taplin, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-319
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Cancer of the prostate; Cancer of prostate; Docetaxel; Carboplatin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Carboplatin

INTERVENTIONS:
Drug: Docetaxel — Given intravenously over 2-3 hours once every three weeks. Participant can continue to receive treatment as long as there is no disease progression or serious side effects.
Drug: Carboplatin — Given intravenously over 2-3 hours once every three weeks. Participant can continue to receive treatment as long as there is no disease progression or serious side effects.

SUMMARY:
The purpose of this study is to look at the effects (good and bad) of the combination of docetaxel and carboplatin for patients who have progressive prostate cancer after chemotherapy with drugs such as docetaxel. The investigators are also studying whether the measurement of two proteins in the blood may predict who will respond to the combination of docetaxel and carboplatin.

DETAILED DESCRIPTION:
Patients will receive both carboplatin and docetaxel. This treatment is given in the outpatient department once every 3 weeks (called one cycle).

One day prior to the day of chemotherapy, patients are given a steroid drug (dexamethasone) to be taken twice a day for 3 days. This helps to decrease the risk of an allergic reaction.

On the day of chemotherapy, both docetaxel and carboplatin will be given through a vein over two to three hours. Docetaxel will be given before carboplatin. In addition, patients receive zofran, an anti-vomiting agent, to try to prevent nausea and vomiting. Study participants are also given a prescription for anti-nausea pills to take at home.

After each cycle of treatment, patients are required to get their bloods checked (between days 8-12 of the cycle). This may be done at an outside laboratory closer to the patient's home.

Treatment will be repeated every three weeks provided the blood tests and physical examination done prior to each treatment are acceptable. If a patient is not able to receive the next scheduled dose of chemotherapy, the doctor will delay the treatment for a week to a maximum of two weeks, beyond which, the patient will be taken off the trial. If there is a delay of more than one week or the study participant has significant side effects, their doctor will decrease the dose of the carboplatin and docetaxel. During the treatment period, doctors may also prescribe medications to treat low red blood cells or low white blood cells.

Before each cycle (every 3 weeks), there will be routine blood tests drawn (about 3 teaspoons) to monitor bone marrow, liver, and kidney functions. These samples will look at two proteins in the blood and may help us predict who will respond to docetaxel and carboplatin. We will also obtain CT scans after every 3 cycles of treatment and at the end of the study. A bone scan will also be done after every 3 cycles if there was evidence of bone involvement on the first bone scan. A bone scan may also be ordered during the study in patients without prior evidence of bone involvement if the doctor suspects that the cancer has now spread to the bone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Evidence of metastatic disease
* Disease progression following androgen deprivation therapy
* Disease progression despite docetaxel-based chemotherapy
* Serum testosterone levels less than 50ng/ml (unless surgically castrated). Patients must continue androgen deprivation with a luteinizing hormone-releasing hormone (LHRH) analogue if they have not undergone orchiectomy.
* No use of antiandrogens for at least 4 weeks
* Cancer and Leukemia Group B (CALGB) performance status less than or equal to 2
* Acceptable white blood cell (WBC), platelets, creatinine and AST counts

Exclusion Criteria:

* Significant peripheral neuropathy defined as grade 2 or higher
* Within 4 weeks since completing external beam radiotherapy or 8 weeks since completing radiopharmaceutical therapy (strontium, samarium)
* Prior platinum-based chemotherapy (cisplatin or carboplatin) for hormone- refractory prostate cancer
* Concomitant chemotherapy, investigational agents or systemic steroids

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-01; Primary Completion 2006-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the efficacy and safety of docetaxel plus carboplatin as salvage chemotherapy in patients with hormone refractory prostate cancer who have progressed on prior docetaxel-based chemotherapy. | 2 years

SECONDARY OUTCOMES:
The secondary objective is to correlate the clinical and prostate-specific antigen (PSA) response with baseline serum chromogranin A (CGA) and neuron-specific enolase (NSE) levels. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Wentworth Douglass Hospital, Dover, New Hampshire
  - Oregon Health and Science University, Portland, Oregon